CLINICAL TRIAL: NCT05722691
Title: Double-Blind, Placebo-Controlled Multicentre Clinical Study for Efficacy and Safety Assessment of the Drug RADAMIN®VIRO for COVID-19 Postexposure Prophylaxis
Brief Title: Study for Efficacy and Safety Assessment of the Drug RADAMIN®VIRO for COVID-19 Postexposure Prophylaxis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAD-012022
Record Dates: First submitted 2023-02-09; First posted 2023-02-10 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; RADAMIN®VIRO; Double-stranded RNA sodium salt
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-stranded RNA sodium salt (Experimental): Arm 1 (n=400) received the study drug RADAMIN®VIRO once intramuscularly, 5 mg (1 vial).
  Interventions: Drug: Double-Stranded RNA sodium salt
- Placebo (Placebo Comparator): Arm 2 (n = 400) received 1 vial of placebo once intramuscularly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Double-Stranded RNA sodium salt — Once intramuscular injection 5 mg (1 vial)
  Other Names: RADAMIN®VIRO
  Arms: Double-stranded RNA sodium salt
Drug: Placebo — Once intramuscular injection (1 vial)
  Arms: Placebo

SUMMARY:
This is Double-Blind, Placebo-Controlled Multicentre Clinical Phase III Study conducted in 10 medical facilities. The objective of the study is to evaluate efficacy and safety of the drug Drug RADAMIN®VIRO, Lyophilisate for Preparation of Solution for Intramuscular and Subcutaneous Administration for COVID-19 Postexposure Prophylaxis

DETAILED DESCRIPTION:
Upon signing the informed consent form and screening, 800 eligible subjects resides with a person with confirmed COVID-19 were randomized at a 1:1 ratio to receive either RADAMIN®VIRO once intramuscularly 5 mg (1 vial) or 1 vial of placebo once intramuscularly

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 80 inclusive (subjects) as of the time of signing the Subject Information Sheet (SIS) Informed Consent Form.
2. A subject resides with a person with confirmed COVID-19 who meets both of the following criteria:

   * The first positive result for SARS-CoV-2 RNA laboratory test with nucleic acid amplification techniques (NAAT) or SARS-CoV-2 antigen with immunochromatographic assay, obtained up to 72 hours prior to randomisation of a subject participating in the study.
   * At least one of the symptoms typical of COVID-19 is observed, with symptoms onset no more than 5 days prior to the randomisation of the subject participating in the study.
3. Negative result for antigen of SARS-CoV-2 with immunochromatographic assay.
4. No symptoms typical of COVID-19 observed.
5. A subject is expected to continue to reside with a person with confirmed COVID-19 during the entire clinical study period; hospitalisation of a person with officially confirmed COVID-19 is not needed at the time of study subject's randomisation.
6. Subject's consent to use reliable contraception methods during the entire study and for 3 weeks after the end of the study. Reliable contraception methods are: sexual abstinence, the use of a condom combined with a spermicidal agent. Female subjects incapable of bearing children (history: hysterectomy, tubal ligation, infertility, menopause for more than 2 years), as well as male subjects with infertility or a history of vasectomy may participate in the study.
7. Availability of SIS Informed Consent Form signed and dated by a patient.
8. Availability of Informed Consent Form for collection of information on COVID-19 signed and dated by a person with confirmed COVID-19.

Exclusion Criteria:

1. Hypersensitivity to the study drug components, procaine.
2. Contraindications to intramuscular injections.
3. Contact with 2 or more persons with confirmed COVID-19 within a month prior to screening or residing with 2 or more people with officially confirmed COVID-19 at the time of screening.
4. Joint residence with more than 10 people.
5. Laboratory-confirmed case of COVID-19 within 6 months prior to randomisation.
6. Vaccination against COVID-19 within less than 4 weeks prior to screening.
7. Use or necessity to use unauthorised pharmaceuticals at the time of screening.
8. Use of immunostimulatory, immunomodulatory, or immunosuppressive medications within 3 months prior to screening.
9. Subjects undergoing renal replacement therapy or with a history of severe renal insufficiency (estimated glomerular filtration rate (GFR) < 30 ml/min/1.73 m2, calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula, within 6 months prior to screening).
10. Primary biliary cirrhosis class C according to the Child - Pugh classification or a history of chronic or active hepatitis B or C.
11. Positive test result for HIV, syphilis, hepatitis B and/or C at the time of screening.
12. Chronic cardiac failure, Functional Class 3 III-IV according to the New York Heart Association (NYHA) Functional Classification.
13. A history of malignant tumours, except for subjects with disease being not observed within the last 5 years, subjects with completely cured basal cell skin cancer, or completely cured carcinoma in situ.
14. Alcohol, pharmacological and/or drug dependence (history and/or at the time of screening).
15. Schizophrenia, schizoaffective disorder, bipolar disorder, or other psychiatric disorder (history or suspected) at the time of screening.
16. Any history data that may complicate, in the opinion of the investigator, interpretation of the study results or create additional risk for the subject due to his/her participation in the study.
17. Unwillingness or inability of a subject to comply with the Protocol procedures (in the opinion of the investigator).
18. Pregnant or lactating women, or women planning a pregnancy.
19. Participation in another clinical study within 3 months prior to enrolment in the present study.
20. Other conditions that prevent the subject from inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Confirmed COVID-19 and presence of at least 1 symptom typical of COVID-19 | From baseline to Visit 3 (days 10-11)
  The number of subjects with confirmed COVID-19 and presence of at least 1 symptom typical of COVID-19

SECONDARY OUTCOMES:
Confirmed COVID-19 and presence of at least 1 symptom typical of COVID-19 | From baseline to Visit 2 (days 3-4), 4 (days 21 ± 1), 5 (days 28 ± 1)
  The number of subjects with confirmed COVID-19 and presence of at least 1 symptom typical of COVID-19
Сonfirmed COVID-19 and absence of symptoms typical for COVID-19 | From baseline to Visit 2 (days 3-4), 3 (days 10-11)
  The number of subjects with confirmed COVID-19 and absence of symptoms typical for COVID-19
Сonfirmed COVID-19 and absence of symptoms typical for COVID-19 | From baseline to Visit 2 (days 3-4), 3 (days 10-11), 4 (days 21 ± 1), 5 (days 28 ± 1)
  The number of subjects with confirmed COVID-19 and absence or presence of symptoms typical of COVID-19
Time to COVID-19 infection | From baseline to Visit 5 (study completion, day 28±1)
  Days to COVID-19 infection
Symptoms typical of COVID-19 | From baseline to Visit 2 (days 3-4), 3 (days 10-11), 4 (days 21 ± 1), 5 (days 28 ± 1)
  The severity of symptoms typical of COVID-19
Duration of symptoms typical of COVID-19 | From baseline to Visit 5 (study completion, day 28±1)
  Duration of symptoms (days) typical of COVID-19
COVID-19 severity evaluation | From baseline to Visit 2 (days 3-4), 3 (days 10-11), 4 (days 21 ± 1), 5 (days 28 ± 1)
  COVID-19 severity evaluation
Hospitalisation due to COVID-19 | From baseline to Visit 5 (study completion, day 28±1)
  The number of subjects who needed hospitalisation due to COVID-19
Total adverse events (AEs) stratified by severity and incidence | From baseline to Visit 5 (study completion, day 28±1)
  Number of AEs stratified by severity and incidence
Incidence of serious adverse events (SAEs), including those due to the use of the study drug/placebo. | From baseline to Visit 5 (study completion, day 28±1)
  Number of SAEs including those due to the use of the study drug/placebo.

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - Regional Budgetary Healthcare Institution Ivanovo Clinical Hospital, Ivanovo
  - Federal State Budgetary Educational Institution of Higher Education Kirov State Medical University of Ministry of Health of the Russian Federation, Kirov
  - State Budgetary Healthcare Institution of Moscow Municipal Clinical Hospital Named after S. I. Spasokukotsky of Moscow Healthcare Department, Moscow
  - Professorskaya Klinika LLC, Perm
  - Avrora MedFort LLC, Saint Petersburg
  - Eco-Safety R&D Centre LLC, Saint Petersburg
  - OrCli Hospital LLC, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education N. P. Ogarev Mordovia State University, Saransk
  - Federal State Budgetary Educational Institution of Higher Education Smolensk State Medical University of Ministry of Health of the Russian Federation Principal Investigator Kozlov Roman Sergeevich, Smolensk
  - Regional State Budgetary Healthcare Institution Clinical Hospital No. 1, Smolensk

IPD SHARING:
Plan to Share IPD: No